CLINICAL TRIAL: NCT06174038
Title: Early Age-Related Hearing Loss Investigation (EARHLI): A Randomized Controlled Trial to Assess the Mechanisms Linking Early Age-Related Hearing Loss and Alzheimer's Disease and Related Dementias
Brief Title: Early Age-Related Hearing Loss Investigation (EARHLI)
Acronym: EARHLI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Aging (NIA) (NIH); University of South Florida (Other); University of Pittsburgh (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Justin S. Golub, Associate Professor of Otolaryngology/Head and Neck Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAU1896; R01AG075083 (NIH)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Hearing Loss; Cognitive Impairment
Keywords: Hearing Loss; Alzheimer's; Alzheimer; Hearing Aid; Memory Loss; Memory; Audiogram; Cognition
MeSH Terms: conditions — Alzheimer Disease; Hearing Loss; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Intervention (Other): Participants will receive 4 sessions across 8 weeks with a later booster session and hearing aid fitting. Each session will take ~75 minutes.
  Interventions: Device: Hearing Intervention
- Health Education Intervention (Other): Participants will receive a modified health education program on healthy aging. It will match the number and length of sessions as the hearing intervention, including compliance/phone checks. Participants will be on a waitlist to obtain hearing aids without fee at the end of their 12-month participation.
  Interventions: Behavioral: Health Education Intervention

INTERVENTIONS:
Device: Hearing Intervention — The hearing intervention includes an auditory needs assessment, hearing aid fitting, establishing Bluetooth connectivity from hearing aids to devices such as smartphones and computers, systematic orientation and instruction in device use, and provision and discussion of hearing "toolkit" materials for self-management and communication strategies. The hearing intervention is person-centered, focusing on identification of individual needs, setting of specific goals, engagement in shared-informed decision-making, and development of self-management abilities. Intervention-centric outcomes (e.g., hearing aid data logging, real ear measures) to verify the best-practices intervention will be gathered at all 5 intervention sessions as well as weeks 16 and 52. Additional visits to troubleshoot hearing aids or address concerns will be scheduled as needed.
  Arms: Hearing Intervention
Behavioral: Health Education Intervention — The evidence-based interactive health education program is designed for older adults and addresses chronic disease and disability prevention. Session content will be individualized for each participant based on a "key," depending on his/her goals/interests. The curriculum includes didactics, activities, and goal setting led by staff trained/certified to deliver the intervention.
  Arms: Health Education Intervention

SUMMARY:
Early Age-Related Hearing Loss Investigation (EARHLI) is a single site study that will randomize late middle age adults to either a hearing intervention (including hearing aids) or a health education intervention. Participants will be followed for 1 year. This study will provide information on reducing cognitive decline in those at risk for Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD).

DETAILED DESCRIPTION:
EARHLI will be a phase II 1:1 randomized controlled trial of a hearing intervention (including prescription hearing aids) versus a health education program. Participants must be 55-75 years old and have early-stage age-related hearing loss and amnestic mild cognitive impairment. The trial will last 1 year and occur at a single site (Columbia University Irving Medical Center). Outcome measurements will include cognition, social engagement, and change in brain organization/connectivity. Assessments will occur at study start, 6 months, and 12 months. A total of 150 participants will be enrolled (75 per intervention group). Participants will also have a hearing test and a blood test. Approximately half of participants will have two MRI scans. As part of participating, all participants will get prescription hearing aids, either at study start or end.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-75 years of age
* Adult-onset hearing loss of approximately mild to moderate in severity (4-frequency 0.5, 1, 2, 4 kHz pure tone average 20 dB to 55 dB HL in better hearing ear)
* Aidable hearing loss, defined by word recognition score in quiet ≥ 60% in better hearing ear
* Amnestic mild cognitive impairment (MCI) defined by Mini-Mental State Exam (MMSE2) score >23, Clinical Dementia Rating (CDR) global score equivalent = 0.5, and ADNI3 criteria of Logical Memory II score of ≤6 if 0-7 years of education, ≤9 if 8-15 years, and ≤11 if ≥16 years
* Availability of a study partner (informant) for the administration of the cognitive screen and the ADCS-Activities of Daily Living-Prevention Instrument (ADCS-ADL-PI)
* Community-dwelling
* Fluent in English or Spanish
* Availability of participant in area for study duration

Exclusion Criteria:

* Self-reported congenital hearing loss, known genetic mutation-related hearing loss, or hearing loss onset before middle age (<45 years old)
* Prior dementia diagnosis
* Reported disability in ≥ 2 activities of daily living (ADLs)
* Current or previous consistent hearing aid user (such as utilization of hearing aids within the past 6 months beyond brief trials)
* Unwillingness to wear hearing aids regularly (≥8 hours/day)
* Medical contraindications to the use of hearing aids (e.g., actively draining ear)
* Corrected vision impairment (worse than 20/63 on MNRead Acuity Chart in worse eye)
* Untreatable conductive hearing loss with air-bone gap > 15 dB in two or more contiguous octave frequencies in both ears

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Free and Cued Selective Reminding Test (FC-SRT) Score | Week 0, Week 28, Week 52
  This is the Cognitive Performance Test # 1 ADCS-PACC 1: Evaluates Episodic Memory. Scoring from 0 - 48 and a higher score translates into a preserved function of the episodic memory.
Delayed Recall Log Memory IIa, (DRLM) Score | Week 0, Week 28, Week 52
  This is the Cognitive Performance Test # 2 ADCS-PACC 2: Evaluates Episodic Memory. Scoring from 0 - 25 and a higher score translates into a preserved function of the episodic memory.
Digit Symbol Substitution Test, (DSST) Score | Week 0, Week 28, Week 52
  This it the Cognitive Performance test # 3 ADCS-PACC 3: Evaluates speed of processing. Scoring from 0 - 91 and a higher score relates to better performance and speed of processing.
Mini-Mental State Examination 2, (MMSE-2) Score | Week 0, Week 28, Week 52
  This is the Cognitive Performance test # 4 ADCS-PACC 4: Evaluates Global Cognition. Scoring from 0 - 30 and a higher score relates to preserved Global Cognition.
Trail Making Test Part B, (TMTB) Score | Week 0, Week 28, Week 52
  This is the Cognitive Performance test # 5 Evaluates Episodic Memory. Scored in terms of the time, in seconds, required to complete the trail. 300 seconds = maximum amount of time. The less seconds it takes to complete the trail, the better performance/ episodic memory.
Activities of Daily Living for Mild Cognitive Impairment, (ADCS-ADLPI) Score | Week 0, Week 28, Week 52
  This is the Cognitive Performance test # 6: Evaluates the ability of patients to perform Activities of Daily Living. Section a. Scored from 0 - 45: Items 1 to 15. Higher score for each activity equals better performance. Section b. Scored from 0 - 5. Item 16 to 20. Higher score equals better performance
Social Activity Frequency | Week 0, Week 28, Week 52
  This is the Social Engagement and Related Socialization test # 1: Evaluates frequency of social activity participation. Participants are asked on a 5-point scale how often during the past 6 months they engaged in 6 common activities involving socialization. A composite score is created
Ability to Participate in Social Roles and Activities (APSR) Score | Week 0, Week 28, Week 52
  This is the Social Engagement and Related Socialization test # 2: Evaluates Social Activity Participation. Scored from 8 - 40 a higher score translates into higher levels of social participation.
Community Integration Measure (CIM) Score | Week 0, Week 28, Week 52
  This is the Social Engagement and Related Socialization test # 3: Evaluates Community Integration/Participation. Scored from 10 - 50. Higher scores indicate higher levels of community integration and participation.
Cohens Social Network Index (SNI) Score | Week 0, Week 28, Week 52
  This is the Social Engagement and Related Socialization test # 4: Evaluates Social Relationships. Scored from 1 - 12. Higher score indicates a larger number of social roles in which the respondent has regular contact.
University of California Loneliness Scale (ULS) Score | Week 0, Week 28, Week 52
  This is the Social Engagement and Related Socialization test # 5: Evaluates Individuals perception of loneliness. The total score ranges from 20 - 80. Higher scores indicate higher loneliness.
Brain MRI Measures | Week 0, Week 52
  Approximately 50% of all participants (random selection) will have a functional brain MRI.

OTHER OUTCOMES:
Hearing Handicap Index for Adults and the Elderly-Short (HHIS) Score | Week 0, Week 28, Week 52
  This test evaluates self perceived hearing handicap. Score ranges from 0 - 48, a higher score indicates higher perception of problems secondary to hearing loss.
Hearing Handicap Index-Short-Significant Other (HHIO) Score | Week 0, Week 28, Week 52
  This test evaluates hearing handicap perceived by subjects significant other. Score ranges from 0 - 48, a higher score indicates higher perception of problems secondary to hearing loss.
Speech, Spatial and Qualities of Hearing Scale (SSQ12) Score | Week 0, Week 28, Week 52
  This test evaluates a range of hearing disabilities across several domains. Scored from 0 - 120, a higher score indicates better hearing.
Vanderbilt Fatigue Scale (VFS) Score | Week 0, Week 28, Week 52
  This test evaluates listening-related fatigue in individuals with hearing loss and other communication-based difficulties. Scored from 0 - 40, a higher score indicates more symptoms of fatigue related to hearing loss.
Pittsburgh Fatigability Scale (PFS) Score | Week 0, Week 28, Week 52
  This test evaluates self-report whole-body physical and mental tiredness related to activities of fixed intensity and duration in adults. Scored from 0 - 50, a higher score indicates more symptoms of fatigue.
Quick Inventory of Depressive Symptoms (QIDS) Score | Week 0, Week 28, Week 52
  Assesses the 9 criterion domains used to diagnose a depressive disorder. Scored 0 - 27 This is the Depression/Depressive Symptom Measure #1: Higher score indicates the presence of more depressive symptoms.
CESD-12 Depression (CES) Score | Week 0, Week 28, Week 52
  This is the Depression/Depressive Symptom Measure # 2: Evaluates symptoms of depression. Possible range of scores is 0 -26, with the higher scores indicating the presence of more symptomatology
RAND Short-Form 36 (SF36) | Week 0, Week 28, Week 52
  This is a general measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Justin S Golub, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Denham MW, Arnold ML, Sanchez VA, Lin FR, Tucker LH, Gomez MC, Fernandez K, Arpi P, Neil H, Boyle S, Selevan S, Sussman TJ, Gmelin T, Fine I, Glynn NW, Teresi J, Noble JM, Goldberg T, Luchsinger JA, Golub JS. Design and Methods of the Early Age-Related Hearing Loss Investigation Randomized Controlled Trial. Otol Neurotol. 2024 Jun 1;45(5):594-601. doi: 10.1097/MAO.0000000000004093. PMID 38728564